CLINICAL TRIAL: NCT00268944
Title: Prospective, Open-label, Single-arm, Exploratory Study of the Effect and Safety of rhGAA in Patients With Advanced Late-onset Pompe Disease Who Are Receiving Respiratory Support
Brief Title: Safety and Effectiveness Study of rhGAA in Patients With Advanced Late-Onset Pompe Disease Receiving Respiratory Support
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU03105
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease (Late-onset); Glycogen Storage Disease Type II (GSD-II); Acid Maltase Deficiency Disease; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg qow
  Other Names: alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The overall objective is to evaluate the safety and efficacy of rhGAA in patients with advanced Late-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged greater than or equal to 18 years
* patient's legally authorized guardian(s) must provide signed, informed consent prior to initiation of study; patient's signature required if patient understands informed consent
* patient must have a documented deficit in acid alpha-glucosidase (GAA) activity , corresponding to the diagnosis of Pompe disease confirmed by documented genotyping
* patient presents with advanced documented symptoms of the disease defined as follows: patient is in a wheel chair and presents diaphragmatic dysfunction and requires invasive ventilation or non invasive ventilation (12 or more hours daily)

Exclusion Criteria:

* patient has received enzyme replacement therapy with GAA from any source
* patient has taken an experimental drug in the 30 days prior to study enrollment, or is currently included in another study involving clinical evaluations; If this is the case, inclusion of the patient in the present study will be subject to prior agreement by Genzyme
* major congenital anomaly
* clinically important organic disease (except for symptoms related to Pompe disease) or any other medical condition, serious intercurrent illness, or other extenuating circumstance that, in the physician's opinion should preclude the patient's participation in the study or may reduce survival
* pregnancy and breastfeeding (women of childbearing age must use a medically accepted method of contraception throughout the entire duration of the trial. Male patients must use a medically accepted birth control method throughout the entire duration of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Treatment effect on muscle strength and functional status. | six months and one year
Treatment effect on pulmonary function and/or ventilation conditions. | six months and one year
Treatment effect on cardiomyopathy noted at inclusion | six months and one year
Treatment effect on fatigue. | six months and one year
Treatment effect on quality of life. | six months and one year
Treatment effect on muscular atrophy. | six months and one year
Overall patient satisfaction with treatment (visual analog scale). | six months and one year
Pharmacodynamics assessment. | six months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Hopital Raymond Poincare, Garches, France